CLINICAL TRIAL: NCT05900141
Title: A Single Arm, Open Label Extension (OLE), Multicenter Study to Evaluate Long-term Safety and Tolerability of Pelacarsen (TQJ230) in Patients With Cardiovascular Disease Who Have Successfully Completed the Apheresis Parent Study.
Brief Title: An Open Label Extension (OLE) Study to Evaluate Long-term Safety and Tolerability of Pelacarsen (TQJ230)
Acronym: OLE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTQJ230A12302E1; 2023-503611-16-00 (Registry Identifier: EUCTR)
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Hyperlipoproteinemia (a)
Keywords: Lipoprotein(a); Cardiovascular disease; Apheresis; Post trial access; pelacarsen (TQJ230)
MeSH Terms: conditions — Hyperlipoproteinemias; Cardiovascular Diseases | interventions — pelacarsen

STUDY DESIGN:
Intervention Model Description: Open-label extension (OLE) study
Masking Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pelacarsen (TQJ230) (Experimental): open-label pelacarsen 80 mg
  Interventions: Drug: Pelacarsen

INTERVENTIONS:
Drug: Pelacarsen — Pelacarsen 80mg s.c. monthly
  Other Names: TQJ230

SUMMARY:
This non-randomized, open-label extension study will provide post-trial access to pelacarsen (TQJ230) to participants in Germany with hyperlipoproteinemia(a) and established cardiovascular disease who have successfully completed the double-blind parent study (CTQJ230A12302).

DETAILED DESCRIPTION:
This study will allow to evaluate a long-term safety and tolerability of pelacarsen (TQJ230) 80 mg QM in patients. All consenting participants from the parent study who meet the eligibility criteria will be participating in this open label extension study. The maximum duration of this study is approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Participant has successfully completed the parent study and is considered safe to participate by Investigator's clinical judgement.

Exclusion Criteria:

* Any medical condition(s) that may put the participant at risk in the investigator's opinion
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, unless they are using effective methods of contraception during dosing and for 16 weeks (= 5 times the terminal half-life) after stopping of study medication

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2028-08-24 (Estimated); Study Completion 2028-08-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events (AEs) or serious adverse events (SAEs), including changes in laboratory evaluations, vital signs qualifying and reported as AEs. | 60 months
  Evaluate long-term safety and tolerability of pelacarsen (TQJ230) in participants with elevated Lp(a) and established cardiovascular disease who have competed the parent study
Duration of drug exposure | 60 months
  Duration of drug exposure will be collected

SECONDARY OUTCOMES:
Number of lipoprotein apheresis sessions performed yearly for year 1, 2, 3, 4 and 5 | 60 months
  Evaluate the long-term effect of pelacarsen on the need for lipoprotein apheresis.
Absolute change in Lp(a) compared to baseline of the parent study. | month 1, month 3, month 6, month 9, month 12, then every 6 months during OLE (up to 60 months)
  Evaluate the long-term effect of pelacarsen on Lp(a) change.
Percentage change in Lp(a) compared to baseline of the parent study. | month 1, month 3, month 6, month 9, month 12, then every 6 months during OLE (up to 60 months)
  Evaluate the long-term effect of pelacarsen on Lp(a) change.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Germany (9):
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cloppenburg
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com